CLINICAL TRIAL: NCT01556984
Title: Changes of Endothelial Function Before and After DSA in Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Xiang Guang-da, Director of Wuhan General Hospital, Wuhan General Hospital of Guangzhou Military Command
Other Study IDs: wz2010007
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes
Keywords: diabetic foot; digital subtraction angiography; endothelial function; Patients with diabetes; Age 40 to 70 years old; Endothelial function are determined
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- DSA group
  Interventions: Other: DSA assay
- control group

INTERVENTIONS:
Other: DSA assay — All patients with diabetic foot perform a DSA assay. Before and after DSA, endothelial function will be measured.
  Groups: DSA group

SUMMARY:
Endothelial dysfunction is the early step of atherosclerosis. Therefore, the investigators hypothesize that digital subtraction angiography (DSA) can damage endothelial function. In this study, the investigators will select 200 diabetic patients who have a DSA for diabetic foot screening. Also, the investigators will select 100 healthy subjects as controls. The endothelial function will be determined by high resolution ultrasound before and after DSA. The investigators will observe the changes of endothelial function after DSA assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic foot
* Age 40 to 70 years old

Exclusion Criteria:

* Heart failure
* Renal failure
* Acute infection

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will select 200 patients with diabetes. DSA will be taken for this group. Endothelial function will be measured before and after DSA. In the meantime, 100 healthy subjects will be selected as controls.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The changes of endothelial function | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China